CLINICAL TRIAL: NCT01364545
Title: Ketogenic Diets for Symptoms of Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Dr Wesley Thevathasan, Honorary consultant neurologist, University of Oxford and the John Radcliffe Hospital, Oxford
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10/H0606/74
Record Dates: First submitted 2011-05-18; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketone ester drink Vs placebo drink (Other): Ketone ester drink Vs placebo drink (cross over study - all patients will recieve both)
  Interventions: Dietary Supplement: Ketone ester drink; Dietary Supplement: Placebo (carbohydrate containing) drink

INTERVENTIONS:
Dietary Supplement: Ketone ester drink — Ketone drink - milligram per kilogram dose, consumed three times daily (at meal times)
Dietary Supplement: Placebo (carbohydrate containing) drink — Placebo drink - containing carbohydrates, matched in calories to ketone, consumed three times daily

SUMMARY:
Parkinson's disease is a progressive condition that harms nerve cells of the brain (neurodegeneration). Current treatments for Parkinson's disease (including levodopa and deep brain stimulation) improve certain symptoms but are not thought to improve the underlying neurodegenerative disease process (they are not a "cure"). The cause of Parkinson's disease is unknown. However, some evidence suggests that tiny structures in the investigators cells called "mitochondria" might be involved. Mitochondria are the powerhouses that produce fuel for the investigators cells. Failure of these 'powerhouses' to supply the energy needs of certain nerve cells might lead to Parkinson's disease. Preliminary evidence suggests that a food called 'ketones' might be able to enhance the function of mitochondria and improve Parkinson's disease symptoms and possibly even the neurodegenerative process. In this study, the investigators would like to investigate this possibility by giving patients with Parkinson's disease dietary supplements of 'ketone esters' in a drink. The investigators will then assess if this improves symptoms of Parkinson's disease.

The study design is a prospective, double blinded, randomised, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Primary Parkinson's disease fulfilling UK Brain Bank criteria
* Age of onset of Parkinson's disease symptoms > 40 years old
* Duration of symptoms over 2 years

Exclusion Criteria:

* Dementia
* Active psychosis
* Deep brain stimulation or apomorphine infusion
* Severe motor fluctuations
* Significant metabolic or uncontrolled medical cormorbidity

Min Age: 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease rating Scale, part III (motor) | 5 days
  Difference between ketone versus placebo scores

SECONDARY OUTCOMES:
Timed motor tasks as per CAPSIT | 5 days
  Hand/Arm movements, 7m walk, 9 hole peg test
Computerised reaction time and cogntive tests | 5 days
  CANTAB
  * SRT and CRT (Task: MOT "Motor screening" practice then RTI "Reaction time")
  * Spatial working memory (Task: SSP "spatial span")
  * Set shifting and visual discrimination (Task: BLC "big circle little circle" practice then IED "intra-extra dimensional shift)
  * Continuous performance task (alertness) (Task: RVP - "Rapid visual processing")
Unified Parkinson's disease rating scale, parts I, II, IV | 5 days
  Difference between ketone versus placebo scores
Dopaminergic medication requirements (expressed as levodopa dose equivalent, mg/day) | 5 days
  Difference between ketone versus placebo doses

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom